CLINICAL TRIAL: NCT04571190
Title: An Adapted Mindfulness-based Stress Reduction Program for Psycho-socially Vulnerable Pregnant Women - a Protocol for a Randomized Feasibility Study in a Danish Hospital-based Outpatient Setting
Brief Title: An Adapted Mindfulness-based Stress Reduction Program for Psycho-socially Vulnerable Pregnant Women.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Copenhagen University Hospital, Hvidovre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 07121971
Record Dates: First submitted 2020-09-18; First posted 2020-09-30 (Actual); Last update posted 2022-05-31 (Actual); Status verified 2020-09

CONDITIONS: Pregnancy, High Risk
Keywords: Prenatal mental health; Pregnancy, High Risk; Mindfulness; Mindfulness-based stress reduction; MBSR; Prenatal mindfulness-based stress reduction
MeSH Terms: interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Intervention Model Description: The design is a single-center feasibility trial comparing prenatal MBSR as add on to usual care with usual care alone. Participants will be randomized in a 1:1 ratio to an intervention or waitlist control group. Participants in the waitlist control group will be offered participation in a MBSR program after a three months follow-up period. Mindfulness training in the control group will thus be initiated postnatal.
Who Masked: Outcomes Assessor
Masking Description: Group affiliation will be concealed for the researcher performing the statistical analyses. Participants will be informed that the overall purpose of the study is to examine the feasibility, acceptability and effect of prenatal MBSR and they are thus not blind to group allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prenatal MBSR (Experimental): The prenatal MBSR program consists of nine two-hour sessions including teachings in mindfulness meditation and yoga. The program is taught by an experienced MBSR instructor with relevant clinical expertise.
  Interventions: Behavioral: Prenatal MBSR
- Usual care (No Intervention): Standard clinical practice, usual care (TAU), imply routine pregnancy visits to the outpatient antenatal clinic at Copenhagen University Hospital, Hvidovre and to a General Practitioner. Usual care include a multidisciplinary approach involving preventive counselling by midwifes, physicians and social workers throughout the pregnancy and follow-up until the early post-partum period.

INTERVENTIONS:
Behavioral: Prenatal MBSR — Prenatal MBSR is an adaptation to the original MBSR program. The essential program elements characterizing MBSR is maintained and integrated with the particular context and specific needs of this group of pregnant women. Adaptations to the MBSR program draw upon both empirical data as well as existing research and theory.
  Other Names: Mindfulness-based stress reduction; MBSR
  Arms: Prenatal MBSR

SUMMARY:
This protocol is for a feasibility study of an adapted mindfulness-based stress reduction (MBSR) program for high-risk pregnant women. The aim is to address the need for more evidence-based options for mental healthcare in pregnancy. MBSR has good evidence in reducing stress, anxiety and depression in both clinical and non-clinical populations, but has not yet been adapted for high-risk pregnancies. The purpose is to evaluate the feasibility, acceptability and potential intervention effects of an adapted MBSR program compared to usual care to inform a randomized controlled trial.

DETAILED DESCRIPTION:
This protocol is for a feasibility study of an adapted mindfulness-based stress reduction (MBSR) program for high-risk pregnant women attending a hospital-based outpatient clinic specialized in antenatal care for high-risk pregnancies. A history of a mental disorder and/or severe psychosocial problems that may pose a risk to the health of the mother and fetus are reasons for referral to the clinic. The protocol is part of the Good start to family life study and the primary aim is to address the need of high-risk pregnant women and care providers for a wider array of evidence-based options to address prenatal mental health care needs. Mindfulness-based interventions are promising interventions for mental disorders with performance equivalent to evidence-based treatments, such as cognitive behavioral therapy and antidepressant medication for some disorders. Moreover, it is an acceptable intervention for pregnant women. A history of any psychopathology or psychosocial adversities, including low social support and abuse, are predictors of mental disorders during and after pregnancy with little diagnostic specificity. Mental disorders or symptoms often continue after birth emphasizing the need for early intervention and prevention. The intention of teaching mindfulness to this group of pregnant women is thus to engage and strengthen their internal resources for optimizing recovery or prevent relapse of mental health disorders during the perinatal period, and to teach skills that may aid the formation of a healthy mother-child relationship.

The objectives of the feasibility study are thus to assess the: (1) acceptance of study participation among at-risk pregnant women; (2) acceptance of allocated interventions; (3) number of referrals to psychiatric treatment during the study period; (4) risk of bias: loss to follow-up in the study arms; acceptance and compliance with the intervention, i.e. attending ≥ 5 sessions; (5) the extent of missing data leading to missing outcomes, and (6) indications of potential intervention effects. The adapted MBSR program will be referred to as prenatal MBSR.

The study is conducted at Copenhagen University Hospital, Hvidovre, Denmark. The design is a single-center feasibility trial comparing prenatal MBSR as add on to usual care with a waitlist control group receiving usual care alone. High-risk pregnant women around 18 weeks gestation (n = 60) will be recruited for the study provided that they are not diagnosed with a major psychiatric illness, psychosis, current substance abuse or suicidality. Participants will be randomized in a1:1 ratio to prenatal MBSR or usual care.

Teaching the skills of mindfulness meditation to a vulnerable group of pregnant women could prove as a viable and non-pharmacological approach to improve mental health and provide support in the transition to parenthood. The outcomes of the feasibility study will inform the design of a fully powered randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Due date no sooner than three months from start of the mindfulness program
* able to speak and write Danish
* available for group intervention scheduled sessions. Being unavailable for two or more sessions is reason for exclusion from study participation.
* written informed consent to study criteria

Exclusion Criteria:

* concurrent substance abuse
* schizophrenia, psychosis, PTSD, schizotypal personality disorder or other major psychiatric disorder
* suicidality

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2021-01-25 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
The Perceived Stress Scale | From baseline to three-months follow-up
  The Perceived Stress Scale 10-item version (PSS-10) is a global measure of the perception of stress. Scores range from 0 - 40 with higher scores pointing to more perceived stress. The Danish consensus version of the PSS-10 can be used in clinical research settings and has good psychometric properties.

SECONDARY OUTCOMES:
The Edinburgh Depression Scale | From baseline to three-months follow-up
  The Edinburgh Depression Scale (EDS) is a widely used screening questionnaire containing questions on how the respondent has felt in the past seven days. Scores range from 0 - 30. A higher score points to more depressive symptoms, and a score of 11 has been suggested as the optimal cut-off for depression according to both DSM-5 and ICD-10 criteria The EDS has been validated as a screening instrument for prenatal and postpartum depression showing good psychometric properties.
The Depression, Anxiety Stress Scales | From baseline to three-months follow-up
  The Depression, Anxiety Stress Scales - 21 (DASS-21) has three subscales designed to discriminate between depression, anxiety and stress in the last week. The DASS excludes somatic items such as sleep disturbance, lack of energy and poor concentration, which may not be valid markers in pregnancy or the postpartum period. Response to each item is rated on a four-point Likert scale ranging from 'never' to 'very much/most of the time'. Scores are calculated for each subscale and higher scores point to more symptoms of stress, anxiety or depression.
WHO-5 | From baseline to three-months follow-up
  The WHO-5 is a short and generic global rating scale measuring subjective well-being. It consists of five statements and the respondent is asked to rate how well each of the statements applies to him or her when considering the last 14 days. Final scores range from 0 - 100 with higher scores representing greater well-being. The scale has adequate validity both as a screening tool for depression and as an outcome measure in clinical trials and has been applied successfully across a wide range of study fields.
Prenatal Reflective functioning | From baselineResponses are rated on a scale from 7 (strongly agree) to 1 (strongly disagree). to three-months follow-up
  Parental reflective functioning refers to the caregiver's capacity to reflect upon his/her own internal mental experiences as well as those of the child. The Prenatal Parental Reflective Functioning Questionnaire (P-PRFQ) is a recently developed 14-item questionnaire for assessing early parental mentalizing capacity. Responses are rated on a scale from 7 (strongly agree) to 1 (strongly disagree). The raw scores range from 14 - 98 and the index sum from 1 - 7. Higher score indicates higher prenatal mentalizing capacity. The P-PRFQ has shown good initial psychometric properties.

OTHER OUTCOMES:
The Experiences Questionnaire: subscale for decentering | From baseline to three-months follow-up
  Decentering reflects the capacity to take a nonjudgmental and accepting stance regarding one´s thoughts and emotions as opposed to identifying with them. The decentering subscale of the experiences questionnaire consists of 11 items with a total score ranging from 11 - 55. Higher scores indicate higher decentering. Initial support has been found for reliability and validity of the scale as a measure of decentering.
The Five Facet Mindfulness Questionnaire | From baseline to three-months follow-up
  The Five Facet Mindfulness Questionnaire (FFMQ) assesses five general facets of being mindful in daily life: observing, describing, acting with awareness, non-reactivity to inner experience, and non-judging of inner experience. Items are rated on a five-point Likert scale ranging from 1 (never or very rarely true) to 5 (very often or always true). Each facet score range from 8 - 40 or from 7 - 35. Higher scores suggest higher levels of mindfulness.
Compassion | From baseline to three-months follow-up
  The Self-Compassion Scale measures the ability to have a healthy stand towards oneself that does not involve evaluations of self-worth. The scale consists of 16 items and responses are given on a 5-point scale from 1 (almost never) to 5 (almost always). Higher scores indicate more self-compassion. The psychometric properties of the scale has been extensive evaluated.

CONTACTS AND LOCATIONS:
Locations (1):
- Copenhagen University Hospital, Amager-Hvidovre, Copenhagen, Capital Region, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stein A, Pearson RM, Goodman SH, Rapa E, Rahman A, McCallum M, Howard LM, Pariante CM. Effects of perinatal mental disorders on the fetus and child. Lancet. 2014 Nov 15;384(9956):1800-19. doi: 10.1016/S0140-6736(14)61277-0. Epub 2014 Nov 14. PMID 25455250
- [Background] Wielgosz J, Goldberg SB, Kral TRA, Dunne JD, Davidson RJ. Mindfulness Meditation and Psychopathology. Annu Rev Clin Psychol. 2019 May 7;15:285-316. doi: 10.1146/annurev-clinpsy-021815-093423. Epub 2018 Dec 10. PMID 30525995
- [Background] Crane RS, Brewer J, Feldman C, Kabat-Zinn J, Santorelli S, Williams JM, Kuyken W. What defines mindfulness-based programs? The warp and the weft. Psychol Med. 2017 Apr;47(6):990-999. doi: 10.1017/S0033291716003317. Epub 2016 Dec 29. PMID 28031068
- [Background] Kuyken W, Warren FC, Taylor RS, Whalley B, Crane C, Bondolfi G, Hayes R, Huijbers M, Ma H, Schweizer S, Segal Z, Speckens A, Teasdale JD, Van Heeringen K, Williams M, Byford S, Byng R, Dalgleish T. Efficacy of Mindfulness-Based Cognitive Therapy in Prevention of Depressive Relapse: An Individual Patient Data Meta-analysis From Randomized Trials. JAMA Psychiatry. 2016 Jun 1;73(6):565-74. doi: 10.1001/jamapsychiatry.2016.0076. PMID 27119968
- [Background] Dhillon A, Sparkes E, Duarte RV. Mindfulness-Based Interventions During Pregnancy: a Systematic Review and Meta-analysis. Mindfulness (N Y). 2017;8(6):1421-1437. doi: 10.1007/s12671-017-0726-x. Epub 2017 Apr 17. PMID 29201244
- [Background] Ludwig DS, Kabat-Zinn J. Mindfulness in medicine. JAMA. 2008 Sep 17;300(11):1350-2. doi: 10.1001/jama.300.11.1350. No abstract available. PMID 18799450
- [Background] Luyten P, Fonagy P. The neurobiology of mentalizing. Personal Disord. 2015 Oct;6(4):366-79. doi: 10.1037/per0000117. PMID 26436580
- [Background] Pajulo M, Tolvanen M, Karlsson L, Halme-Chowdhury E, Ost C, Luyten P, Mayes L, Karlsson H. THE PRENATAL PARENTAL REFLECTIVE FUNCTIONING QUESTIONNAIRE: EXPLORING FACTOR STRUCTURE AND CONSTRUCT VALIDITY OF A NEW MEASURE IN THE FINN BRAIN BIRTH COHORT PILOT STUDY. Infant Ment Health J. 2015 Jul-Aug;36(4):399-414. doi: 10.1002/imhj.21523. Epub 2015 Jun 19. PMID 26096692
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Cox JL, Holden JM, Sagovsky R. Detection of postnatal depression. Development of the 10-item Edinburgh Postnatal Depression Scale. Br J Psychiatry. 1987 Jun;150:782-6. doi: 10.1192/bjp.150.6.782. PMID 3651732
- [Background] Smith-Nielsen J, Matthey S, Lange T, Vaever MS. Validation of the Edinburgh Postnatal Depression Scale against both DSM-5 and ICD-10 diagnostic criteria for depression. BMC Psychiatry. 2018 Dec 20;18(1):393. doi: 10.1186/s12888-018-1965-7. PMID 30572867
- [Background] Lovibond PF, Lovibond SH. The structure of negative emotional states: comparison of the Depression Anxiety Stress Scales (DASS) with the Beck Depression and Anxiety Inventories. Behav Res Ther. 1995 Mar;33(3):335-43. doi: 10.1016/0005-7967(94)00075-u. PMID 7726811
- [Background] Lee D. The convergent, discriminant, and nomological validity of the Depression Anxiety Stress Scales-21 (DASS-21). J Affect Disord. 2019 Dec 1;259:136-142. doi: 10.1016/j.jad.2019.06.036. Epub 2019 Jun 30. PMID 31445339
- [Background] Topp CW, Ostergaard SD, Sondergaard S, Bech P. The WHO-5 Well-Being Index: a systematic review of the literature. Psychother Psychosom. 2015;84(3):167-76. doi: 10.1159/000376585. Epub 2015 Mar 28. PMID 25831962
- [Background] Fonagy P, Luyten P, Moulton-Perkins A, Lee YW, Warren F, Howard S, Ghinai R, Fearon P, Lowyck B. Development and Validation of a Self-Report Measure of Mentalizing: The Reflective Functioning Questionnaire. PLoS One. 2016 Jul 8;11(7):e0158678. doi: 10.1371/journal.pone.0158678. eCollection 2016. PMID 27392018
- [Background] Fresco DM, Moore MT, van Dulmen MH, Segal ZV, Ma SH, Teasdale JD, Williams JM. Initial psychometric properties of the experiences questionnaire: validation of a self-report measure of decentering. Behav Ther. 2007 Sep;38(3):234-46. doi: 10.1016/j.beth.2006.08.003. Epub 2007 Apr 24. PMID 17697849
- [Background] Baer RA, Smith GT, Lykins E, Button D, Krietemeyer J, Sauer S, Walsh E, Duggan D, Williams JM. Construct validity of the five facet mindfulness questionnaire in meditating and nonmeditating samples. Assessment. 2008 Sep;15(3):329-42. doi: 10.1177/1073191107313003. Epub 2008 Feb 29. PMID 18310597
- [Background] Pommier E, Neff KD, Toth-Kiraly I. The Development and Validation of the Compassion Scale. Assessment. 2020 Jan;27(1):21-39. doi: 10.1177/1073191119874108. Epub 2019 Sep 13. PMID 31516024
- [Background] Billingham SA, Whitehead AL, Julious SA. An audit of sample sizes for pilot and feasibility trials being undertaken in the United Kingdom registered in the United Kingdom Clinical Research Network database. BMC Med Res Methodol. 2013 Aug 20;13:104. doi: 10.1186/1471-2288-13-104. PMID 23961782
- [Background] Eldridge SM, Chan CL, Campbell MJ, Bond CM, Hopewell S, Thabane L, Lancaster GA; PAFS consensus group. CONSORT 2010 statement: extension to randomised pilot and feasibility trials. Pilot Feasibility Stud. 2016 Oct 21;2:64. doi: 10.1186/s40814-016-0105-8. eCollection 2016. PMID 27965879
- [Derived] Skovbjerg S, Kolls M, Kjaerbye-Thygesen A, Fjorback LO. Mindfulness-Based Stress Reduction adapted to pregnant women with psychosocial vulnerabilities - a randomized feasibility trial in a Danish hospital-based outpatient setting. Pilot Feasibility Stud. 2025 Jun 21;11(1):86. doi: 10.1186/s40814-025-01670-0. PMID 40544301
- [Derived] Skovbjerg S, Birk D, Bruggisser S, Wolf ALA, Fjorback L. Mindfulness-based stress reduction adapted to pregnant women with psychosocial vulnerabilities-a protocol for a randomized feasibility study in a Danish hospital-based outpatient setting. Pilot Feasibility Stud. 2021 Jun 3;7(1):118. doi: 10.1186/s40814-021-00860-w. PMID 34082839